CLINICAL TRIAL: NCT01724294
Title: Non-interventional, Post-marketing Study to Evaluate the Correlation Between Clinical and Biological Factors and IPI as Prognostic Factors in Patients With DLBCL in First Line Treatment With R-CHOP
Brief Title: An Observational Study of MabThera/Rituxan (Rituximab) in Combination With CHOP Chemotherapy in First-Line in Patients With Diffuse Large B-Cell Lymphoma
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28497
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, observational study will evaluate the correlation between clinical and biological factors and International Prognostic Index (IPI) as prognostic factors in patients with diffuse large B-cell lymphoma receiving first-line treatment with MabThera/Rituxan (rituximab) in combination with CHOP chemotherapy. Eligible patients receiving treatment according to standard of care and local guidelines will be followed for the duration of treatment (approximately 8 months) and during 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >18 years of age
* Patients with diagnosed diffuse large B-cell lymphoma in first-line treatment with R-CHOP

Exclusion Criteria:

* Prior chemotherapy treatment for diffuse large B-cell lymphoma
* Contra-indications or exclusion criteria according to the Summary of Product Characteristics for MabThera/Rituxan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diffuse large B-cell lymphoma treated in first line with R-CHOP
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2012-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Treatment patterns in clinical practice: Number of treatment cycles received | approximately 4 years

SECONDARY OUTCOMES:
Event-free survival | approximately 4 years
Response rates | approximately 4 years
Safety: Incidence of adverse events | approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bucharest, Romania